CLINICAL TRIAL: NCT00092053
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Persistence of the Effect of Oral Monthly Ibandronate on Bone Reception in Postmenopausal Women in Osteoporosis
Brief Title: Study of Investigational Drug in Osteoporosis (MK-0217-908)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0217-908
Record Dates: First submitted 2004-09-21; First posted 2004-09-24 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Postmenopausal; Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Ibandronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive 3 placebo tablets once a month, for 3 months, on the first day of each treatment cycle.
  Interventions: Drug: Placebo
- ibandronate 100 mg (Experimental): Participants will receive 2 ibandronate 50 mg tablets and 1 placebo tablet once a month, for 3 months, on the first day of each treatment cycle.
  Interventions: Drug: ibandronate
- ibandronate 150 mg (Experimental): Participants will receive 3 ibandronate 50 mg tablets once a month, for 3 months, on the first day of each treatment cycle.
  Interventions: Drug: ibandronate

INTERVENTIONS:
Drug: Placebo — tablets
  Arms: Placebo
Drug: ibandronate — 50 mg tablets
  Arms: ibandronate 100 mg; ibandronate 150 mg

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of an investigational drug in postmenopausal women with osteoporosis. The primary hypothesis of this study is that in postmenopausal women with osteoporosis, oral monthly ibandronate, at doses of 100 mg and 150 mg, does not achieve persistence in reduction of bone resorption throughout the monthly dosing interval, as demonstrated by a larger change in the serum carboxyterminal crosslinked telopeptide of Type I collagen (CTX-I) log-transformed fraction from baseline four weeks post dose compared to one week post dose, during the third month of treatment, in the participants taking ibandronate than in the participants taking placebo.

ELIGIBILITY:
Inclusion Criteria: -postmenopausal for at least 3 years, with osteoporosis at any of the following sites: [BMD > 2.0 standard deviations below young normal mean bone mass for the hip trochanter, PA lumbar spine (L1 to L4), total hip, or femoral neck based on the normative database provided by each individual manufacturer].

* willing to take study-supplied calcium and vitamin D supplement (or equivalent) and to discontinue any non-study calcium supplements for run-in period and the duration of the study. Exclusion Criteria: -pregnant or lactating, or of childbearing potential.
* participated in another therapeutic trial with an investigational compound within 30 days of randomization.
* history of hypersensitivity to any component of ibandronate tablets or has hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
* an abnormality of the esophagus which delays esophageal emptying such as stricture or achalasia.
* unable to stand or sit upright for at least 60 minutes once a month.
* current use of illicit drugs, or history of drug or alcohol abuse within the past five years.
* has any of the following: hypocalcemia; any severe malabsorption syndrome; moderate or severe hypertension which is uncontrolled; new onset angina or myocardial infarction within six months of entry into the study; evidence for impaired renal function; organ transplantation; or other significant end organ diseases (genitourinary, cardiovascular, endocrine, hepatic, psychiatric, renal, hematologic, or pulmonary).
* history of or evidence of metabolic bone disease (other than postmenopausal bone loss).
* clinical fracture in the past year.
* is receiving or has received treatment prior to randomization which might influence bone turnover.
* is receiving or expected to receive during the course of the study any medication (other than study medication) which might alter bone or calcium metabolism, including Vitamin A in excess of 10,000 IU per day or Vitamin D in excess of 5000 IU per day, calcitonin, phenytoin, heparin, or lithium.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2004-12; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Change in serum levels of CTX-I (log-transformed fraction) from Week 9 to Week 12 | Baseline, Week 9, Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC